CLINICAL TRIAL: NCT01193361
Title: A Phase 2A Study of BMS-791325 in Combination With Peg Interferon Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment-Naïve Subjects With Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Ph IIA Study (SOC +/- NS5B)
Acronym: HEPCAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI443-012
Record Dates: First submitted 2010-08-25; First posted 2010-09-01 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 - BMS-791325 plus peg-interferon alfa-2a and ribavirin (Experimental)
  Interventions: Drug: BMS-791325; Drug: Peg-interferon alfa-2a; Drug: Ribavirin
- Arm 2 - BMS-791325 plus peg-interferon alfa-2a and ribavirin (Experimental)
  Interventions: Drug: BMS-791325; Drug: Peg-interferon alfa-2a; Drug: Ribavirin
- Arm 3 - Placebo plus peg-interferon alfa-2a and ribavirin (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Peg-interferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-791325 — Tablets, Oral, 75 mg, twice daily, 4-48 weeks depending on response
  Arms: Arm 1 - BMS-791325 plus peg-interferon alfa-2a and ribavirin
Drug: BMS-791325 — Tablets, Oral, 150 mg, twice daily, 4-48 weeks depending on response
  Arms: Arm 2 - BMS-791325 plus peg-interferon alfa-2a and ribavirin
Drug: Placebo — Tablets, Oral, 0 mg, twice daily, 4-48 weeks depending on response
  Arms: Arm 3 - Placebo plus peg-interferon alfa-2a and ribavirin
Drug: Peg-interferon alfa-2a — Syringe, Subcutaneous Injection, 180 µg, once weekly, 4-48 weeks depending on response
  Other Names: Pegasys
Drug: Ribavirin — Tablets, Oral, 1000 or 1200 mg based on weight, twice daily, 4-48 weeks depending on response
  Other Names: Copegus

SUMMARY:
At least 1 dose of BMS-791325 can be identified which is safe, well tolerated, and efficacious when combined with peg-interferon alfa-2a (pegIFNα-2a)/ribavirin (RBV) for the treatment of treatment-naïve, chronically-infected hepatitis C virus (HCV) genotype 1 subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects chronically infected with HCV genotype 1 as documented by: positive for anti-HCV antibody, HCV RNA, or a positive HCV genotype test at least 6 months prior to Screening, and positive for HCV RNA and anti-HCV antibody at Screening
* HCV RNA ≥ 10*5* IU/mL at Screening
* Less than 4 weeks total prior therapy with an IFN formulation (ie, IFNα, pegIFNα-2a), or RBV and no exposure to IFN or RBV within 24 weeks of Randomization
* Results of a biopsy obtained ≤ 24 months prior to Randomization showing no evidence of cirrhosis
* Body Mass Index (BMI) of 18 to 35 kg/m², inclusive. BMI = weight (kg)/ [height (m)]² at Screening

Exclusion Criteria:

* Liver transplant recipients
* Documented or suspected HCC by imaging or liver biopsy
* Evidence of a medical condition associated with chronic liver disease other than HCV (such as but not limited to: hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History of chronic hepatitis B virus (HBV) as documented by HBV serologies (eg. HBsAg-seropositive). Patients with resolved HBV infection may participate (eg. HBsAb-seropositive)
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety, as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Formal analysis at week 4 (and upon occurrence)
Safety, as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Formal analysis at week 12 (and upon occurrence)
Safety, as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Formal analysis at week 24 post treatment (and upon occurrence)
Safety, as measured by the frequency of serious adverse events (SAEs) and discontinuations due to adverse events (AEs) | Formal analysis at week 48 post treatment (and upon occurrence)
Antiviral activity, as determined by the proportion subjects with eRVR | Week 4
Antiviral activity, as determined by the proportion subjects with eRVR | Week 12

SECONDARY OUTCOMES:
Proportion of subjects with rapid virologic response (RVR), defined as undetectable HCV RNA | Week 4
Proportion of subjects with complete early virologic response (cEVR), defined as undetectable HCV RNA | Week 12
Proportions of subjects with a 12-week SVR (SVR12) and 24-week SVR (SVR24), defined as undetectable HCV RNA at off treatment follow-up | Week 12
Proportions of subjects with a 12-week SVR (SVR12) and 24-week SVR (SVR24), defined as undetectable HCV RNA at off treatment follow-up | Week 24
Resistant HCV variants associated with virologic failure | End of treatment (Week 48) or upon early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (10):
  - Advanced Clinical Research Institute, Anaheim, California
  - Loyola University Medical Center, Maywood, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, P.A., Baltimore, Maryland
  - Claudia T. Martorell, Md, Llc, Springfield, Massachusetts
  - Charlotte Gastroenterology & Hepatology, Pllc, Charlotte, North Carolina
  - Options Health Research, Llc, Tulsa, Oklahoma
  - The North Texas Research Institute, Arlington, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx